CLINICAL TRIAL: NCT00076921
Title: Research on China Tobacco Control Epidemiology and Intervention
Brief Title: Epidemiology & Intervention Research for Tobacco Control
Status: Completed | Type: Observational
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Frances Stillman, Associate Professor, Johns Hopkins Bloomberg School of Public Health
Other Study IDs: 1209; 5R01HL073699 (NIH)
Record Dates: First submitted 2004-02-06; First posted 2004-02-09 (Estimated); Last update posted 2013-04-10 (Estimated); Status verified 2013-04

CONDITIONS: Lung Diseases
MeSH Terms: conditions — Lung Diseases

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Biospecimen Retention: None Retained — No bio-specimens collected. Sampled nicotine from buildings only.
Oversight: Data Monitoring Committee: No

SUMMARY:
To characterize the development of tobacco control capacity with staff from the Chinese Center's for Disease control (CDCs) at the provincial level and to have them develop and implement population-level interventions to build awareness and knowledge concerning the harms of smoking that could help lead to policy action being taken to protect the population from the harms caused by smoking. Compare capacity, policy and, second-hand smoke exposure and smoking rates in selected provinces to national levels.

DETAILED DESCRIPTION:
China is a particularly critical country for global tobacco control. It has the world's largest number of smokers, approximately 350 million, and the immense market afforded by the 60 percent of men who smoke and the 95 percent of women who do not smoke represents a prize target for the multinational tobacco companies. China has ratified the Framework Convention for Tobacco Control (FCTC) and now needs to implement its provisions across a large and diverse population. In this application, we propose a program of evidence-based community interventions to be implemented at the province and local levels with the overall objective of developing an approach for implementation nationally.

This application builds on a long-standing partnership between the Chinese Center for Disease Control and Prevention (China CDC), the Peking Union Medical College (PUMC) and the Johns Hopkins Bloomberg School of Public Health. That partnership began in 1995 with an agreement to collaborate on the conduct of China's 1996 national smoking survey. Our principal collaborator over those years, Dr. Gong-Huan Yang, is now Deputy Director of the China CDC and responsible for tobacco control at the national level. In the four years of funding to date from the Fogarty International Center (FIC), we have carried out a project in selected communities in three provinces, including urban and rural areas that provide a foundation for the intervention approach in this proposal. Specifically, we have carried out quantitative and qualitative studies to assess barriers to tobacco control and readiness for interventions, measured levels of airborne nicotine in key public environments, and developed capacity-building approaches. Our original FIC supported study involved three countries, China, Mexico and Brazil. However, this application will focus solely on China, as the latter two countries developed the necessary infrastructure and capacity to conduct research, publish their research findings, and seek further grants and government funding to sustain progress.

This application proposes a tobacco control study that will involve 7 provinces in a CDC-led initiative to develop a systematic mix of approaches. The plan uses strategies based on experiences from our work in China and from the American Stop Smoking Intervention Study for Cancer Prevention (ASSIST) and anticipates barriers that have been identified in the data collected to date. In the intervention provinces, the China CDC will team with the provincial-level CDCs to assess capacity for tobacco control and the current status of tobacco control, using an adapted version of the Strength of Tobacco Control (SOTC) index developed for evaluating ASSIST. This systematic characterization will highlight capacity needs. An extensive capacity development program, based in distance-based methods, will be used. We have the overall objective of preparing the China CDC to implement a proven approach to tobacco control at the national level. A household survey will be conducted and compared to the national survey results. Second-hand smoking will be assessed in selected locations in the 7 provinces.

ELIGIBILITY:
No eligibility criteria

Ages: 15 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Household representatives in 7 selected provinces will complete a survey.
Sampling Method: Probability Sample
Enrollment: 15705 (Actual)
Dates: Start 2002-09; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Compare smoking rates and second-hand smoke exposure in 7 provinces to national data. | 3 years
  A national household survey was conducted. Provincial household surveys that adapted questions from the national survey were administered to gain provincial estimates.

SECONDARY OUTCOMES:
Change or increase in number of tobacco control policies at the provincial level | 3 years
  Policies in hospital, schools, worksites, government buildings, transportation facilities will be assessed to determine if they have implemented a policy.
Determine change in ability to conduct tobacco control strategies. | 3 years.
  An assessment of the provinces ability or capacity to conduct tobacco control strategies were compared at baseline and at the end of the project.

CONTACTS AND LOCATIONS:
Overall Officials: Frances Stillman, Principal Investigator — Johns Hopkins University

REFERENCES:
- [Background] Stillman FA, Wipfli HL, Lando HA, Leischow S, Samet JM. Building capacity for international tobacco control research: the global tobacco research network. Am J Public Health. 2005 Jun;95(6):965-8. doi: 10.2105/AJPH.2004.047183. PMID 15914817